CLINICAL TRIAL: NCT01224275
Title: Group Based Care Versus Individual Care- Effects on Parents Satisfaction and Health
Brief Title: Group Based Care Versus Individual Care
Acronym: GBAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ewa Andersson, Dr., Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2007/553
Record Dates: First submitted 2010-10-19; First posted 2010-10-20 (Estimated); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Patient Satisfaction
Keywords: group based care; antenatal care; parents satisfaction; Antenatal care´s organization and patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group antenatal care (Experimental): The first arm is midwife which allocated to group based antenatal care. They have education in this model of care and follow up meeting to secure the intervention
  Interventions: Other: group based care
- Individual antenaal care (No Intervention): the second arm include midwife which allocated to traditional care as control group.

INTERVENTIONS:
Other: group based care — Midwives is randomized and allocated to group based antenatal care. The midwives have a manual for the model of care.
  Other Names: intervention including midwifes in the care.
  Arms: Group antenatal care

SUMMARY:
The Study compares group based care versus individual given care-effects on patient satisfaction and health. Midwives will be randomized to either traditional antenatal care (Individual care) or group based antenatal care(intervention).

DETAILED DESCRIPTION:
In the RCT the midwife is randomized.There are a multicenter study. Before the study started the midwives received education about the study. Then they randomized with simple randomization per site(clinics). The midwives also have follow up meeting with the research team during the recruting period. The parents are informed about the study at the booking appointment, after that they can choose if they want to participate in the study and are allocated to either intervention or control, based on the woman's date of birth. The main aim is to investigate parents' satisfaction of antenatal group based care. The RCT is based on three questionnaires which both women and their partners receive, the first at baseline before they receive different models of care, and the second questionnaire distributed four to six months after birth and the last one year after birth. Descriptive and inferential statistics will be used in the analysis.A power calculation is made and the study schould have a total number of 350 partners.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to Speak Swedish

Exclusion Criteria:

* Non speaking Swedish

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1150 (Actual)
Dates: Start 2008-08; Primary Completion 2014-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Group based antenatal care versus Individual care- parent´s satisfaction with care | 6 years
  Satisfaction with care and involvement of partner, three questionnaire to parents in control group and intervention group, which measure the satisfaction with care

SECONDARY OUTCOMES:
socialization with other parents | 4 years
  The study include this secondary outcome, measure with two qustionnarie four to six mounts after birth and the second qustionnarie one year after birth. The questionnare to borth group(conrtil group and intervention griup)
Self reported health effect on mother and child | 6 years
  Measure the health with instrument as EPDS scale and question regarding health, parental stress and breastfeeding.Four to six months and one year after birth.
  The questionnaire is sending out to both woman and partner.

CONTACTS AND LOCATIONS:
Overall Officials: Eva andersson, Dr, Principal Investigator — eva andersson
Locations (1):
- Karolinska Institut-Woman and childrens health, Stockholm, Sweden